CLINICAL TRIAL: NCT03411343
Title: A Randomized Comparison Between Interscalene and Costoclavicular Infraclavicular Brachial Plexus Blocks For Arthroscopic Shoulder Surgery
Brief Title: Interscalene Block Versus Costoclavicular Block for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Clinical Instructor, Department of Anesthesia, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 889/17
Record Dates: First submitted 2018-01-05; First posted 2018-01-26 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Pain, Postoperative; Shoulder Pain; Surgical Procedure, Unspecified; Diaphragmatic Paralysis
Keywords: Postoperative Shoulder Analgesia; Hemidiaphragmatic Paralysis; Alternative blocks
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain; Respiratory Paralysis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene Block (Active Comparator): Patients randomized to receive an intesrcalene block.
  Interventions: Procedure: Interscalene Block
- Costoclavicular Infraclavicular Block (Experimental): Patients randomized to receive a costoclavicular infraclavicular block.
  Interventions: Procedure: Costoclavicular Infraclavicular Block

INTERVENTIONS:
Procedure: Interscalene Block — Injection with ultrasound guidance of 20mL of levobupivacaine 0.5% with 5 micrograms of epinephrine per mL in the interscalene groove of the brachial plexus.
  Arms: Interscalene Block
Procedure: Costoclavicular Infraclavicular Block — Ultrasound guided brachial plexus block injecting 20mL of 0.5% levobupivacaine with 5 micrograms of epinephrine per mL in between the cords of the brachial plexus at the costoclavicular infraclavicular space.
  Arms: Costoclavicular Infraclavicular Block

SUMMARY:
Interscalene brachial plexus block constitutes the analgesic criterion standard for shoulder surgery. However, it is associated with a high incidence of hemidiaphragmatic paralysis (HDP) that may not be tolerated by patients with chronic pulmonary disease. This randomized controlled trial (RCT) will compare ultrasound-guided interscalene block (ISB) and costoclavicular infraclavicular block (CCICB) in patients undergoing arthroscopic shoulder surgery.

The main outcome is static pain at 30 minutes after arrival in the post anesthesia care unit (PACU) as measured by a numerical rate scale (NRS) from 0 to 10. Our research hypothesis is that interscalene and costoclavicular infraclavicular blocks will result in equivalent postoperative analgesia at 30 minutes in the PACU. The equivalence margin is set at 2 points.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing arthroscopic shoulder surgery
* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy
* Coagulopathy
* Obstructive or restrictive pulmonary disease
* Renal failure
* Hepatic failure
* Allergy to local anesthetics
* Pregnancy
* Prior surgery in the corresponding side of the neck or infraclavicular fossa
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Static pain at 30 minutes after arrival in the PACU | 30 minutes
  Evaluated with a NRS from 0 to 10

SECONDARY OUTCOMES:
Static pain at 60 minutes after arrival in the PACU | 60 minutes
  Evaluated with a NRS from 0 to 10
Postoperative static pain at 2 hours | 2 hours
  Evaluated with a NRS from 0 to 10
Postoperative static pain at 3 hours | 3 hours
  Evaluated with a NRS from 0 to 10
Postoperative static pain at 6 hours | 6 hours
  Evaluated with a NRS from 0 to 10
Postoperative static pain at 12 hours | 12 hours
  Evaluated with a NRS from 0 to 10
Postoperative static pain at 24 hours | 24 hours
  Evaluated with a NRS from 0 to 10
Incidence of HDP at 30 minutes after interscalene or costoclavicular infraclavicular block | 30 minutes post injection
  Ultrasound diagnosed HDP
Incidence of HDP at 30 minutes after arrival to PACU | 30 minutes after arrival to the PACU
  Ultrasound diagnosed HDP
Block performance time | 1 hour before surgery
  Time from skin disinfection until the end of local anesthetic injection
Sensory and Motor block score | 30 minutes post injection
  Sensorimotor block assessed every 5 minutes until 30 minutes using a 8-point composite score
Incidence of complete block | 30 minutes post injection
  Percentage of blocks with a minimal sensorimotor composite score of 6 points out of a maximum of 8 points at 30 minutes post injection
Procedural pain during blocks | 1 hour before surgery
  Evaluated with a NRS from 0 to 10
Onset time | 1 hour before surgery
  Time required to reach a minimal sensorimotor composite score of 6 points out of a maximum of 8 points
Intraoperative opioid requirements | Intraoperative period
  Total amount of fentanyl required during general anesthesia
Surgical duration | Intraoperative period
  Time between skin incision and closure
Postoperative opioid consumption | 24 hours after surgery
  Total amount of morphine required during the first 24 hours after surgery
Patient satisfaction | 24 hours after surgery
  Patient satisfaction measured using a NRS 0 to 10 (0 = unsatisfied; 10 =very satisfied)
Block- and opioid-related side effects | 1 week
  Incidence of side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Martinez J, Sala-Blanch X, Ramos I, Gomar C. Combined infraclavicular plexus block with suprascapular nerve block for humeral head surgery in a patient with respiratory failure: an alternative approach. Anesthesiology. 2003 Mar;98(3):784-5. doi: 10.1097/00000542-200303000-00031. No abstract available. PMID 12606927
- [Background] Aliste J, Bravo D, Finlayson RJ, Tran DQ. A randomized comparison between interscalene and combined infraclavicular-suprascapular blocks for arthroscopic shoulder surgery. Can J Anaesth. 2018 Mar;65(3):280-287. doi: 10.1007/s12630-017-1048-0. Epub 2017 Dec 19. PMID 29270914
- [Background] Leurcharusmee P, Elgueta MF, Tiyaprasertkul W, Sotthisopha T, Samerchua A, Gordon A, Aliste J, Finlayson RJ, Tran DQH. A randomized comparison between costoclavicular and paracoracoid ultrasound-guided infraclavicular block for upper limb surgery. Can J Anaesth. 2017 Jun;64(6):617-625. doi: 10.1007/s12630-017-0842-z. Epub 2017 Feb 15. PMID 28205117
- [Background] Lloyd T, Tang YM, Benson MD, King S. Diaphragmatic paralysis: the use of M mode ultrasound for diagnosis in adults. Spinal Cord. 2006 Aug;44(8):505-8. doi: 10.1038/sj.sc.3101889. Epub 2005 Dec 6. PMID 16331304
- [Background] Tran DQ, Dugani S, Finlayson RJ. A randomized comparison between ultrasound-guided and landmark-based superficial cervical plexus block. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):539-43. doi: 10.1097/AAP.0b013e3181faa11c. PMID 20975470
- [Background] Karmakar MK, Sala-Blanch X, Songthamwat B, Tsui BC. Benefits of the costoclavicular space for ultrasound-guided infraclavicular brachial plexus block: description of a costoclavicular approach. Reg Anesth Pain Med. 2015 May-Jun;40(3):287-8. doi: 10.1097/AAP.0000000000000232. No abstract available. PMID 25899958
- [Background] Spence BC, Beach ML, Gallagher JD, Sites BD. Ultrasound-guided interscalene blocks: understanding where to inject the local anaesthetic. Anaesthesia. 2011 Jun;66(6):509-14. doi: 10.1111/j.1365-2044.2011.06712.x. PMID 21568985
- [Background] Flohr-Madsen S, Ytrebo LM, Valen K, Wilsgaard T, Klaastad O. A randomised placebo-controlled trial examining the effect on hand supination after the addition of a suprascapular nerve block to infraclavicular brachial plexus blockade. Anaesthesia. 2016 Aug;71(8):938-47. doi: 10.1111/anae.13504. PMID 27396247
- [Background] Tashjian RZ, Deloach J, Porucznik CA, Powell AP. Minimal clinically important differences (MCID) and patient acceptable symptomatic state (PASS) for visual analog scales (VAS) measuring pain in patients treated for rotator cuff disease. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):927-32. doi: 10.1016/j.jse.2009.03.021. Epub 2009 Jun 16. PMID 19535272
- [Derived] Aliste J, Bravo D, Layera S, Fernandez D, Jara A, Maccioni C, Infante C, Finlayson RJ, Tran DQ. Randomized comparison between interscalene and costoclavicular blocks for arthroscopic shoulder surgery. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-100055. doi: 10.1136/rapm-2018-100055. Online ahead of print. PMID 30635497